CLINICAL TRIAL: NCT02892331
Title: The High Intensity Exercise to Promote Accelerated Improvements in CardiorEspiratory Fitness (HI-PACE) Study
Brief Title: Effects of Exercise Training Intensity on Fitness and Insulin Sensitivity in African Americans
Acronym: HI-PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Damon Swift, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R03DK105297-01A1 (NIH)
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Insulin Resistance; Sedentary Lifestyle
Keywords: exercise; insulin resistance; mitochondrial function; arterial stiffness; exercise intensity; fitness
MeSH Terms: conditions — Obesity; Insulin Resistance; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): This group does not change physical activity during the intervention period, but will receive exercise training after the study is complete
- MOD-INT (Experimental): The Moderate intensity exercise training (MOD-INT) group will exercise at a moderate aerobic exercise intensity for 24 weeks
  Interventions: Behavioral: Moderate intensity exercise training (MOD-INT)
- HIGH-INT (Experimental): High Intensity exercise training (HI-INT) group will exercise at a high aerobic intensity for 24 weeks
  Interventions: Behavioral: High Intensity exercise training (HI-INT)

INTERVENTIONS:
Behavioral: Moderate intensity exercise training (MOD-INT) — Participants in the MOD-INT group will exercise at the heart rate associated with 45-55% VO2 max. The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)
  Arms: MOD-INT
Behavioral: High Intensity exercise training (HI-INT) — Participants in the HI-INT group will exercise at the heart rate associated with 70-80% VO2 max (heart rate ranges will be updated at mid-intervention CRF assessment). The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)3
  Arms: HIGH-INT

SUMMARY:
African Americans are at a substantially greater type 2 diabetes risk compared to Caucasians; however, very little data are available on the effects of exercise training on type 2 diabetes risk factors in at risk African Americans. The present proposal will evaluate the effects of 6 months of moderate versus vigorous intensity aerobic exercise training on fitness, insulin sensitivity, mitochondrial capacity, skeletal muscle oxidative/insulin sensitivity markers, adiposity, and quality of life in African Americans.

DETAILED DESCRIPTION:
African Americans have a much greater risk of type 2 diabetes compared to Caucasians in the United States. Similarly, recent evidence has emerged that fitness level, a major risk factor for type 2 diabetes also tends to be lower in African Americans. Many scientific studies have shown that exercise training has a beneficial impact on fitness levels and a variety of other type 2 diabetes risk factors such as the reduction of glucose/insulin levels, and body fat Importantly, studies performed in mostly Caucasian populations suggest that exercise training at a vigorous intensity may promote greater improvements in type 2 diabetes risk factors compared to moderate intensity exercise, which may suggest that it has greater promise in reducing type 2 diabetes risk. However, few exercise training studies compare the health benefits of different exercise training programs (such as exercise intensity) in African Americans, which is clinically important due to their greater type 2 diabetes risk, and that fact that they are less likely to meet public health recommendations for physical activity compared to their Caucasian counterparts.

The High Intensity exercise to Promote Accelerated improvements in CardiorEspiratory fitness (HI-PACE) study will evaluate the effect of exercise intensity on cardiorespiratory fitness (CRF) and insulin sensitivity in obese (BMI: 30-45) African Americans (40-65 yrs.) with at least 1 additional T2D risk factor. Participants (n=60) will be recruited in collaboration with the ECU Center for Health Disparities, and subsequently randomized to moderate intensity (MOD-INT, n=20) or high intensity (HIGH-INT, n=20) aerobic exercise training, or to a control group (CON, n=20) for 24 weeks. Supervised exercise training will be performed at a heart rate associated with ~50% and ~75% of VO2 max in the MOD-INT and the HIGH-INT groups, respectively at the same exercise volume of 600 MET-minutes per week (consistent with public health recommendations). The primary outcome is the change in CRF, which will be assessed at baseline, mid-intervention, and follow-up. Insulin sensitivity will be measured via an intravenous glucose tolerance test at baseline and follow-up. Other secondary measures include mitochondrial oxidative capacity using infrared and measurements on muscle biopsies (PGC-1α and other indices of mitochondrial content), the expression of a protein involved with insulin action (GLUT-4 expression) in skeletal muscle as well as systemic inflammation, adiposity, quality of life and exercise enjoyment measures.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Body mass index 30-45 kg/m2
* sedentary/low active (step count ≤ 6,500 step/day)
* capable and willing to give written informed consent and understand exclusion criteria
* willingness to accept group assignment from randomization
* No resistance training and no structured aerobic exercise for > 20 minutes per day, 3+ days per week, for the last 6 months
* conditions that are contraindicated for exercise training

Exclusion Criteria:

* Resting blood pressure > 180 mm Hg systolic and/or >100 mm Hg diastolic; individuals on blood pressure medications meeting the blood pressure criteria are eligible
* Diagnosis of type 1 or 2 diabetes, and/or fasting glucose >125 mg/dL
* Medication for the treatment of type 1 or type 2 diabetes
* Bariatric surgery including gastric banding or bypass (potential effects on energy intake)
* Factors that may limit adherence to intervention or affect conduct of the trial
* Unable or unwilling to communicate with staff
* Failure to complete run-in or baseline testing
* Hospitalization for depression or severe mental illness in the last 6 months
* Not physically capable of performing the exercise required of the study protocol
* Consuming more than 14 alcoholic beverages per week
* Plan to be away from the Pitt County area more than 3 weeks in the next 3 months
* Lack support from a primary health care provider or family members
* Significant weight loss in the past year (> 20 pounds) or are currently using weight loss medications.
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Another member of the household who is currently a participant or staff member of this study
* Other temporary intervening event, such as sick spouse, or bereavement
* Other medical, psychiatric, or behavioral limitations that may interfere with study participation or the ability to follow the intervention protocol
* Underlying diseases or conditions likely to limit lifespan and/or affect the safety of the intervention
* Cancer requiring treatment in the past 5 years with anything but excellent prognosis
* Self-reported HIV, tuberculosis, Hepatitis B, or Hepatitis C
* History or evidence of serious arrhythmias, cardiomyopathy, congestive heart failure, aortic aneurism, myocardial infarction or heart transplantation
* Renal disease: urine protein > 100 mg/dl, serum creatinine ≥ 1.5 mg/dl or currently receiving dialysis.
* Auto-immune diseases (such as Lupus, Multiple Sclerosis, Graves' disease, or Rheumatoid arthritis)
* Chronic obstructive lung disease, peripheral vascular disease or angina that limits ability to follow exercise protocol
* History of stroke or transient ischemic attack
* History of vascular aneurysms
* History of bleeding disorders
* Pregnancy or plans to become pregnant
* Dieting or plans to diet, or in a weight loss program
* Any other medical condition or disease that is life threatening or that can interfere with or be aggravated by exercise.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-10; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damon L Swift, Ph.D., Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGee JE, Barefoot SG, Gniewek NR, Brophy PM, Clark A, Dubis GS, Ryan TE, Houmard JA, Vos P, Raedeke TD, Swift DL. High-intensity exercise to promote accelerated improvements in cardiorespiratory fitness (HI-PACE): study protocol for a randomized controlled trial. Trials. 2019 Aug 8;20(1):484. doi: 10.1186/s13063-019-3611-1. PMID 31395096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The HI-PACE study was conducted in Greenville, NC at East Carolina University. Participants were recruited from the local Greenville, NC and Pitt County areas. Methods of recruitment included sending information to mailing list of local agencies, working with community partners, the ECU health disparity center, social media advertisements and local newspaper advertisements. Recruitment for the study began in Fall of 2016
Pre-assignment Details: individuals interested in study participation came in for a screening visit to determine initial eligibility. After this, those that remained eligible, did a "run-in" period where they wore an accelerometer for 7 consecutive days. When they returned with their accelerometer, a blood draw was performed for screening labs. After this, participants were scheduled for primary and secondary outcome measures. After completion of these outcomes measures, they were randomized to study groups.
Groups:
- Control (CON): This group does not change physical activity during the intervention period, but will receive exercise training after the study is complete
- Moderate Intensity Training (MOD-INT): The Moderate intensity exercise training (MOD-INT) group will exercise at a moderate aerobic exercise intensity for 24 weeks
  Moderate intensity exercise training (MOD-INT): Participants in the MOD-INT group will exercise at the heart rate associated with 45-55% VO2 max. The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)
- High Intensity Training (HIGH-INT): High Intensity exercise training (HI-INT) group will exercise at a high aerobic intensity for 24 weeks
  High Intensity exercise training (HI-INT): Participants in the HI-INT group will exercise at the heart rate associated with 70-80% VO2 max (heart rate ranges will be updated at mid-intervention CRF assessment). The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)3
Period: Overall Study
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Started | 18 | 16 | 18
Completed | 16 | 13 | 14
Not Completed | 2 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Sick family member | 0 | 0 | 1
Not completed — Corona virus pandemic | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Blood pressure was too elevated | 0 | 1 | 0
Not completed — participant did not disclose she had an excluded medical condition and was disenrolled | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate Intensity (MOD-INT): The Moderate intensity exercise training (MOD-INT) group will exercise at a moderate aerobic exercise intensity for 24 weeks
  Moderate intensity exercise training (MOD-INT): Participants in the MOD-INT group will exercise at the heart rate associated with 45-55% VO2 max. The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)
- High Intensity Exercise (HIGH-INT): High Intensity exercise training (HI-INT) group will exercise at a high aerobic intensity for 24 weeks
  High Intensity exercise training (HI-INT): Participants in the HI-INT group will exercise at the heart rate associated with 70-80% VO2 max (heart rate ranges will be updated at mid-intervention CRF assessment). The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)3
- Total: Total of all reporting groups
Arm/Group | Control (CON) | Moderate Intensity (MOD-INT) | High Intensity Exercise (HIGH-INT) | Total
Number analyzed (Participants) | 18 | 16 | 18 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 18 | 52
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (7.1) | 50.2 (7.6) | 48.0 (8.0) | 49.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 16 | 43
  Male | 4 | 3 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 18 | 16 | 18 | 52
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 18 | 52
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index is calculated by dividing the participants' weight in kilograms by height in meters squared
  kg/m^2 | 32.9 (6.2) | 35.6 (4.8) | 36.8 (5.8) | 35.1 (5.8)
Weight [Mean (Standard Deviation); unit: kg] — Weight was taken on scale in a hospital gown
  kg | 90.7 (17.0) | 98.7 (13.6) | 104.9 (20.7) | 98.1 (18.2)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was taken after a 5 minute rest in the seated position
  mmHg | 128.5 (13.6) | 129.8 (10.8) | 133.9 (12.6) | 130.8 (12.6)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — diastolic blood pressure was measured in the seated position after a 5 minute rest
  mmHg | 81.8 (10.9) | 83.1 (9.6) | 85.1 (8.8) | 83.3 (9.7)
Cardiorespiratory fitness (L/min) [Mean (Standard Deviation); unit: L/min] — Cardiorespiratory fitness was measured as the maximal level of oxygen consumed during a treadmill exercise test
  L/min | 2.0 (0.6) | 1.8 (0.4) | 2.0 (0.6) | 1.9 (0.5)
Cardiorespiratory fitness (mL/kg/min) [Mean (Standard Deviation); unit: mL/kg/min] — Cardiorespiratory fitness is measured as the maximal amount of O2 that body consumes during a maximal exercise test. This value is adjusted by the participant's body weight
  mL/kg/min | 21.6 (6.0) | 18.5 (4.3) | 18.7 (3.8) | 19.5 (4.9)
Glucose [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of glucose in the blood from a fasting blood sample
  mg/dL | 93.3 (10.5) | 93.2 (6.9) | 94.5 (11.6) | 93.7 (9.9)
Insulin [Mean (Standard Deviation); unit: ulU/mL] — Describes the concentration of insulin in a fasted blood sample
  ulU/mL | 13.6 (8.0) | 15.4 (9.3) | 16.4 (8.2) | 15.1 (8.4)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of cholesterol from a fasting blood sample
  mg/dL | 185.6 (26.7) | 177.3 (40.5) | 166.4 (33.2) | 176.4 (33.8)
Low density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 111.3 (27.5) | 107.3 (40.5) | 98.4 (28.8) | 105.6 (32.1)
High density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 54.7 (15.6) | 53.9 (13.6) | 48.3 (14.3) | 52.2 (14.6)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — The concentration of triglycerides from a fasting blood sample
  mg/dL | 97.7 (46.1) | 80.0 (23.2) | 98.1 (40.2) | 92.6 (38.6)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] — C-reactive protein is a marker of inflammation and is measured from a fasting blood sample
  mg/L | 5.5 (4.4) | 5.6 (4.9) | 6.1 (7.8) | 5.7 (5.9)
Pulse wave velocity [Mean (Standard Deviation); unit: m/sec] — Pulse wave velocity is a measure of arterial stiffness
  m/sec | 7.4 (1.1) | 6.9 (1.3) | 7.6 (1.2) | 7.3 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiorespiratory Fitness
Description: Fitness will be measured using a modified Balke protocol on a treadmill. Participants will walk at an initial speed of 2.0 mph with 0% grade for the first 3 minutes after which the treadmill speed will increase to 3.0 mph for the next 3 minutes. The treadmill grade will be increased by 2.5% every 3 minutes until volitional exhaustion. Maximal oxygen consumption (Liters of O2 per minute) will be measured using a True Max 2400 Metabolic Measurement Cart (Parvomedics, Salt Lake City Utah).
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters of oxygen/min
Groups:
- Moderate Intensity Exercise (MOD-INT): The Moderate intensity exercise training (MOD-INT) group will exercise at a moderate aerobic exercise intensity for 24 weeks
  Moderate intensity exercise training (MOD-INT): Participants in the MOD-INT group will exercise at the heart rate associated with 45-55% VO2 max. The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)
- High Intensity Exercise HIGH-INT: High Intensity exercise training (HI-INT) group will exercise at a high aerobic intensity for 24 weeks
  High Intensity exercise training (HI-INT): Participants in the HI-INT group will exercise at the heart rate associated with 70-80% VO2 max (heart rate ranges will be updated at mid-intervention CRF assessment). The exercise volume will be 600 MET-minutes per week, which is consistent with current public health guidelines (500-1,000 MET-minutes)3
Arm/Group | Control (CON) | Moderate Intensity Exercise (MOD-INT) | High Intensity Exercise HIGH-INT
Number analyzed (Participants) | 16 | 13 | 13
Liters of oxygen/min | -0.15 [-0.32 to 0.03] | 0.12 [-0.07 to 0.31] | 0.22 [0.03 to 0.41]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Exercise HIGH-INT; Comparison between the CON and the HIGH-INT group; Test type: Superiority; p = 0.006, ANCOVA — VO2 testing was not performed for one participant in the HIGH-INT group
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Exercise (MOD-INT); Comparison between the CON and MOD-INT group; Test type: Superiority; p = 0.045, ANCOVA — VO2 testing was not performed for one participant in the HIGH-INT group
Statistical Analysis 3: Comparison: Moderate Intensity Exercise (MOD-INT) vs High Intensity Exercise HIGH-INT; Comparison between MOD-INT and High-INT groups; Test type: Superiority — VO2 testing was not performed for one participant in the HIGH-INT group; p = 0.449, ANCOVA

2. Secondary Outcome: Change in Body Fat Percentage
Description: Dual-energy X-ray absorptiometry will be used to measure changes in body fat percentage
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of body fat
Arm/Group | Control | MOD-INT | HIGH-INT
Number analyzed (Participants) | 16 | 13 | 13
percentage of body fat | 0.09 [-0.89 to 1.07] | -0.26 [-1.35 to 0.83] | -0.71 [-1.80 to 0.38]
Statistical Analysis 1: Comparison: Control vs HIGH-INT; Comparison between the CON and High-INT groups; Test type: Superiority; p = 0.276, ANCOVA
Statistical Analysis 2: Comparison: Control vs MOD-INT; Comparison between the CON and MOD-INT groups; Test type: Superiority; p = 0.633, ANCOVA
Statistical Analysis 3: Comparison: MOD-INT vs HIGH-INT; Comparison between the MOD-INT and HIGH-INT groups; Test type: Superiority; p = 0.555, ANCOVA

3. Secondary Outcome: Change in Body Weight
Description: Weight will be measured using a calibrated scale. Weight will be measured in kg
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 13 | 14
kg | 0.87 [-1.04 to 2.8] | -0.37 [-2.45 to 1.70] | -0.42 [-2.52 to 1.67]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON group and the HIGH-INT group; Test type: Superiority; p = 0.370, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and the MOD-INT group; Test type: Superiority; p = 0.383, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison for the MOD-INT and HIGH-INT groups; Test type: Superiority; p = 0.0972, ANCOVA

4. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference will be measured at the natural waist (midway between the inferior border of the rib cage and the superior aspect of the iliac crest) with a Gulick tape measure. Both landmarks (the inferior border of the ribcage and the superior aspect of the iliac crest) will be marked and the distance will be measured to determine the appropriate measurement site. Staff will confirm that: 1) the measurement tape remains horizontal; 2) the tape touches the entire circumference of the participant; 3) abdominal tissue is not compressed; 3) the tape measure is not within abdominal folds; 4) the measurement is taken at the end of normal respiration. The measurement will be repeated an additional time, and the reported value will be the average of these measurements. Both measurements must be within 0.5 cm to be considered acceptable for data purposes.
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 13 | 13
cm | -1.42 [-3.9 to 1.0] | 0.41 [-2.2 to 3.0] | -1.3 [-4.0 to 1.5]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and the HIGH-INT groups; Test type: Superiority; p = 0.932, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and MOD-INT groups; Test type: Superiority; p = 0.307, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT and the HIGH-INT groups; Test type: Superiority; p = 0.376, ANCOVA

5. Secondary Outcome: Change in Low Density Lipoprotein
Description: Low density lipoprotein will be measured from a fasting blood sample
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 12 | 13
mg/dL | -7.1 [-15.2 to 1.1] | -0.12 [-9.53 to 9.3] | 2.3 [-6.9 to 11.5]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and the HIGH-INT groups; Test type: Superiority; p = 0.136, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and the MOD-INT group; Test type: Superiority; p = 0.262, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT group and the HIGH-INT groups; Test type: Superiority; p = 0.715, ANCOVA

6. Secondary Outcome: Change in High Density Lipoprotein
Description: High density lipoprotein will be measured from a fasted blood sample
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 12 | 13
mg/dL | -3.4 [-6.7 to -0.17] | -1.1 [-4.9 to 2.7] | 1.3 [-2.3 to 5.0]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and High-INT groups; Test type: Superiority; p = 0.056, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and MOD-INT groups; Test type: Superiority; p = 0.349, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT and HIGH-INT groups; Test type: Superiority; p = 0.359, ANCOVA

7. Secondary Outcome: Changes in Total Cholesterol
Description: Total Cholesterol will be measured in a fasting blood sample
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 12 | 13
mg/dL | -10.4 [-20.5 to -0.21] | -0.21 [-12.3 to 11.8] | -0.71 [-12.5 to 11.1]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and HIGH-INT groups; Test type: Superiority; p = 0.224, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and MOD-INT groups; Test type: Superiority; p = 0.199, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT and the HIGH-INT groups; Test type: Superiority; p = 0.952, ANCOVA

8. Secondary Outcome: Change in Triglycerides
Description: Triglyceride levels will be measured from a fasting blood sample
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 12 | 13
mg/dL | -10.9 [-22.4 to 0.58] | 4.0 [-9.5 to 17.6] | -13.3 [-26.1 to -0.45]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and HIGH-INT groups; Test type: Superiority; p = 0.783, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and MOD-INT groups; Test type: Superiority; p = 0.098, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD and HIGH-INT groups; Test type: Superiority; p = 0.071, ANCOVA

9. Secondary Outcome: Change in Systemic Inflammation
Description: High sensitivity c-reactive protein will be measured at baseline and follow-up
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 14 | 11 | 13
mg/L | 0.142 [-3.11 to 3.39] | 0.159 [-3.54 to 3.84] | 0.31 [-3.09 to 3.73]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and the HIGH-INT groups; Test type: Superiority; p = 0.940, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and MOD-INT groups; Test type: Superiority; p = 0.994, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT and HIGH-INT groups; Test type: Superiority; p = 0.940, ANCOVA

10. Secondary Outcome: Change in Fasting Glucose
Description: Fasting glucose will be measured from a fasting blood sample
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 12 | 13
mg/dL | -2.81 [-6.7 to 1.1] | -2.5 [-6.6 to 2.5] | -2.0 [-6.3 to 2.4]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison of the CON and HIGH-INT groups; Test type: Superiority; p = 0.769, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison of the CON and MOD-INT groups; Test type: Superiority; p = 0.800, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Test type: Superiority; p = 0.769, ANCOVA

11. Secondary Outcome: Change in Insulin
Description: Fasting insulin value will be measured from a blood sample
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: ulU/mL
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 12 | 13
ulU/mL | -2.68 [-6.4 to 1.0] | -2.69 [-6.9 to 1.6] | -2.7 [-6.8 to 1.4]
Statistical Analysis 1: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and the MOD groups; Test type: Superiority; p = 1.000, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison of HIGH-INT and CON groups; Test type: Superiority; p = 0.993, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT and the HIGH-INT groups; Test type: Superiority; p = 0.994, ANCOVA

12. Secondary Outcome: Change in Insulin Sensitivity
Description: Insulin sensitivity will be measured using an intravenous glucose tolerance test
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: (mu/l)^-1.min^-1
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 11 | 6 | 7
(mu/l)^-1.min^-1 | 0.60 [-0.53 to 1.74] | 0.59 [-0.94 to 2.12] | 0.44 [-1.02 to 1.83]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in insulin sensitivity (CON vs. HIGH-INT); Test type: Superiority; p = 0.821, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in insulin sensitivity (CON vs. MOD-INT); Test type: Superiority; p = 0.985, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in insulin sensitivity (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.856, ANCOVA

13. Secondary Outcome: Change in Arterial Stiffness
Description: Arterial stiffness will be measured using pulse wave velocity.
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: m/sec
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 13 | 11 | 12
m/sec | -0.21 [-0.76 to 0.34] | 0.68 [0.08 to 1.28] | 0.47 [-0.11 to 1.04]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison between the CON and HIGH-INT groups; Test type: Superiority; p = 0.093, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Comparison between the CON and the MOD-INT groups; Test type: Superiority; p = 0.033, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Comparison between the MOD-INT and HIGH-INT groups; Test type: Superiority; p = 0.602, ANCOVA

14. Secondary Outcome: Change in Mitochondrial Enzymes
Description: Mitochondrial enzymes (citrate synthase, pgc1aplha and complex1-5)
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: U/mU
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 9 | 9 | 9
U/mU
  PGC1 alpha | -0.17 [-0.45 to 0.09] | 0.02 [-0.26 to 0.30] | -0.02 [-0.1 to 0.30]
  Citrate synthase | -0.01 [-0.18 to 0.16] | 0.02 [-0.14 to 0.18] | 0.17 [0.00 to 0.34]
  Complex 1 | -0.36 [-0.96 to 0.24] | 0.17 [-0.43 to 0.77] | -0.05 [-0.65 to 0.56]
  Complex 2 | -0.06 [-0.49 to 0.36] | 0.16 [-0.30 to 0.61] | -0.05 [-0.48 to 0.38]
  Complex 3 | 0.07 [-0.19 to 0.34] | 0.09 [-0.19 to 0.37] | -0.01 [-0.26 to 0.24]
  Complex 4 | -0.32 [-0.80 to 0.58] | 0.23 [-0.22 to 0.67] | 0.01 [-0.41 to 0.43]
  Complex 5 | -0.05 [-0.19 to 0.10] | 0.01 [-0.07 to 0.27] | 0.01 [-0.14 to 0.16]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in PGC1A (CON vs. HIGH-INT); Test type: Superiority; p = 0.424, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in PGC1A (CON vs. MOD-INT); Test type: Superiority; p = 0.308, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in PGC1a (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.844, ANCOVA
Statistical Analysis 4: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in citrate synthase (CON vs. HIGH-INT); Test type: Superiority; p = 0.135, ANCOVA
Statistical Analysis 5: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in Citrate synthase (CON vs. MOD-INT); Test type: Superiority; p = 0.800, ANCOVA
Statistical Analysis 6: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in citrate synthase; Test type: Superiority; p = 0.195, ANCOVA
Statistical Analysis 7: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in complex I; Test type: Superiority; p = 0.459, ANCOVA
Statistical Analysis 8: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in complex 1 (CON vs. MOD-INT groups); Test type: Superiority; p = 0.213, ANCOVA
Statistical Analysis 9: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in complex II (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.971, ANCOVA
Statistical Analysis 10: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in complex III (CON vs. HIGH-INT); Test type: Superiority; p = 0.634, ANCOVA
Statistical Analysis 11: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in Complex III (CON vs. MOD-INT groups); Test type: Superiority; p = 0.919, ANCOVA
Statistical Analysis 12: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in complex III; Test type: Superiority; p = 0.574, ANCOVA
Statistical Analysis 13: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in Complex IV (CON vs. HIGH-INT); Test type: Superiority; p = 0.295, ANCOVA
Statistical Analysis 14: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in complex IV (CON vs. MOD-INT); Test type: Superiority; p = 0.097, ANCOVA
Statistical Analysis 15: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in complex IV; Test type: Superiority; p = 0.468, ANCOVA
Statistical Analysis 16: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in complex V; Test type: Superiority; p = 0.589, ANCOVA
Statistical Analysis 17: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in complex V (CON vs. MOD-INT); Test type: Superiority; p = 0.196, ANCOVA
Statistical Analysis 18: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in Complex V (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.436, ANCOVA

15. Secondary Outcome: Change in Quality of Life
Description: Quality of life (QOL) will be measured by the short form health survey (SF-36). SF36 consists of 36 questions that measure patient's HRQoL in 8 domains: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH) that represent the physical HRQoL, vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH) that represent the mental HRQoL. Each domain is scored from 0 (worst health status) to 100 (best health status).
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 16 | 13 | 13
score on a scale
  General Health | -1.6 [-4.0 to 0.8] | 1.3 [-1.4 to 3.9] | -1.0 [-3.7 to 1.62]
  Physical health | -0.18 [-3.5 to 3.1] | 0.57 [-3.1 to 4.2] | 2.4 [-1.2 to 6.1]
  Role Physical | -0.22 [-3.2 to 2.8] | -1.2 [-4.5 to 2.2] | 1.1 [-2.2 to 4.4]
  Bodily pain | -3.6 [-8.1 to 0.9] | -2.1 [-7.0 to 2.9] | 0.2 [-4.8 to 5.3]
  Vitality | 1.1 [-1.7 to 3.9] | -1.51 [-4.5 to 1.5] | 2.6 [-0.4 to 5.7]
  Social Function | -0.15 [-3.6 to 3.3] | -5.2 [-9.0 to -1.3] | 0.7 [-3.2 to 4.6]
  Mental health | 0.8 [-1.6 to 3.1] | -2.2 [-4.8 to 0.4] | 0.65 [-1.9 to 3.3]
  Role Emotional | 0.8 [-1.5 to 3.1] | -0.0 [-2.5 to 2.5] | 2.3 [-0.2 to 4.9]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison of general health subscale (CON vs. HIGH INT); Test type: Superiority; p = 0.756, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); General Health Subscale (CON vs. MOD-INT); Test type: Superiority; p = 0.115, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); General Health Subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.225, ANCOVA
Statistical Analysis 4: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Physical health Sub-scale (CON vs. HIGH-INT); Test type: Superiority; p = 0.758, ANCOVA
Statistical Analysis 5: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Physical health subscale (CON vs. MOD-INT); Test type: Superiority; p = 0.759, ANCOVA
Statistical Analysis 6: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Physical Health subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.465, ANCOVA
Statistical Analysis 7: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Role Physical subscale (CON vs. HIGH-INT); Test type: Superiority; p = 0.549, ANCOVA
Statistical Analysis 8: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Role Physical Subscale (CON vs. MOD-INT); Test type: Superiority; p = 0.679, ANCOVA
Statistical Analysis 9: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Role Physical Subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.334, ANCOVA
Statistical Analysis 10: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Bodily pain subscale (CON vs. HIGH-INT); Test type: Superiority; p = 0.273, ANCOVA
Statistical Analysis 11: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Bodily pain subscale (CON vs. MOD-INT); Test type: Superiority; p = 0.642, ANCOVA
Statistical Analysis 12: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Bodily Pain Subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.520, ANCOVA
Statistical Analysis 13: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Vitality subscale (CON vs. HIGH-INT); Test type: Superiority; p = 0.460, ANCOVA
Statistical Analysis 14: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Vitality sub-scale (CON vs. MOD-INT group); Test type: Superiority; p = 0.203, ANCOVA
Statistical Analysis 15: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Vitality subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.058, ANCOVA
Statistical Analysis 16: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Social Function subscale (CON vs. HIGH-INT); Test type: Superiority; p = 0.739, ANCOVA
Statistical Analysis 17: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Social Function subscale (CON vs. MOD-INT); Test type: Superiority; p = 0.059, ANCOVA
Statistical Analysis 18: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Social Function sub-scale (HIGH-INT vs. MOD-INT); Test type: Superiority; p = 0.0380, ANCOVA
Statistical Analysis 19: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Comparison of mental health subscale (CON vs. HIGH-INT); Test type: Superiority; p = 0.950, ANCOVA
Statistical Analysis 20: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in mental health subscale (CON Vs. MOD INT); Test type: Superiority; p = 0.096, ANCOVA
Statistical Analysis 21: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in mental health subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.127, ANCOVA
Statistical Analysis 22: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in role emotional subscale (CON vs HIGH-INT); Test type: Superiority; p = 0.373, ANCOVA
Statistical Analysis 23: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in role emotional sub-scale; Test type: Superiority; p = 0.630, ANCOVA
Statistical Analysis 24: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in role emotional subscale (MOD vs. HIGH-INT); Test type: Superiority; p = 0.034, ANCOVA
Statistical Analysis 25: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in role emotional subscale (CON vs. MOD-INT); Test type: Superiority; p = 0.070, ANCOVA
Statistical Analysis 26: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in physical health sub-scale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.945, ANCOVA

16. Secondary Outcome: Change in Quality of Life (Mental Health and Physical Health Summary Scores)
Description: The SF-36 also produces a measure of overall physical health (physical component score [PCS]) and overall mental health (mental component score [MCS]). Scoring of these items are standardized using means and standard deviations from the general US population. Aggregate PCS and MCS scores are standardized using a linear T-Score transformation to have a mean of 50 and a standard deviation of 10. A higher score indicates better quality of life and a lower score indicates worsened quality of life.
Time Frame: Baseline to 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control (CON) | Moderate Intensity Exercise (MOD-INT) | High Intensity Exercise HIGH-INT
Number analyzed (Participants) | 16 | 13 | 13
score on a scale
  Mental health (sum) | 0.75 [-1.7 to 3.3] | -2.7 [-5.4 to 0.09] | 1.6 [-1.2 to 4.4]
  Physical health (sum) | -2.02 [-4.6 to 0.6] | 0.02 [-2.8 to 2.9] | -0.11 [-3.0 to 2.8]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Exercise HIGH-INT; Change in the mental health sum scale (CON vs. HIGH-INT); Test type: Superiority; p = 0.650, ANCOVA
Statistical Analysis 2: Comparison: Moderate Intensity Exercise (MOD-INT) vs High Intensity Exercise HIGH-INT; Change in mental health (sum) subscale (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.034, ANCOVA
Statistical Analysis 3: Comparison: Control (CON) vs High Intensity Exercise HIGH-INT; Change in physical health (sum); Test type: Superiority; p = 0.330, ANCOVA
Statistical Analysis 4: Comparison: Control (CON) vs Moderate Intensity Exercise (MOD-INT); Change in physical health (sum) subscale; Test type: Superiority; p = 0.297, ANCOVA

17. Secondary Outcome: Changes in Physical Activity Levels
Description: Participants will wear an ActivPal accelerometer for seven consecutive days, 24-hrs/day. The change in steps will be be evaluated from baseline to 24 weeks
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 10 | 9 | 9
steps per day | 604.2 [-792.9 to 2001.3] | 2311.0 [817.9 to 3804.1] | 2242.3 [763.3 to 3721.4]
Statistical Analysis 1: Comparison: Control (CON) vs High Intensity Training (HIGH-INT); Change in steps (CON vs. HIGH-INT); Test type: Superiority; p = 0.109, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Moderate Intensity Training (MOD-INT); Change in steps (CON vs. MOD-INT); Test type: Superiority; p = 0.099, ANCOVA
Statistical Analysis 3: Comparison: Moderate Intensity Training (MOD-INT) vs High Intensity Training (HIGH-INT); Change in steps (MOD-INT vs. HIGH-INT); Test type: Superiority; p = 0.947, ANCOVA

18. Secondary Outcome: Change in Dietary Composition
Description: Food Frequency Questionnaire (FFQ) contains approximately 105 items grouped by categories and is completed for both frequency of consumption as well as portion size selections by the individual. The questionnaire, upon completion, provides estimated daily intake values for selected nutrients (kilocalories, macronutrients, and micronutrients) and provides information on food group servings.
Time Frame: Baseline and 24 weeks
Population: Error in processing the data and it was lost
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks per participants
Arm/Group | Control (CON) | Moderate Intensity Training (MOD-INT) | High Intensity Training (HIGH-INT)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 1/16 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (CON) (N=18) | Moderate Intensity Training (MOD-INT) (N=16) | High Intensity Training (HIGH-INT) (N=18)
Elevated blood pressure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Participant had elevated blood pressure after randomization that was higher than the trend noted in pre-randomization visits

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02892331/Prot_SAP_000.pdf